CLINICAL TRIAL: NCT04591392
Title: Evaluation of the Safety and Efficacy of the reSept ASD Occluder to Treat Patients With Clinically Significant Secundum Atrial Septal Defect
Brief Title: Safety and Efficacy Study of reSept ASD Occluder for Treating Secundum ASD
Acronym: ASCENT ASD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: atHeart Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008-022
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Heart Septal Defect; Heart Septal Defects, Atrial; Heart Defects, Congenital; Cardiovascular Abnormalities; Cardiovascular Diseases; Heart Diseases; Congenital Abnormalities
MeSH Terms: conditions — Heart Septal Defects; Heart Septal Defects, Atrial; Heart Defects, Congenital; Cardiovascular Abnormalities; Cardiovascular Diseases; Heart Diseases; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Device (Experimental): ASD closure with the reSept ASD Occluder
  Interventions: Device: reSept ASD Occluder

INTERVENTIONS:
Device: reSept ASD Occluder — Transcatheter closure of secundum ASD using a permanent implant

SUMMARY:
Evaluation of the safety and efficacy of the reSept ASD Occluder to treat patients with clinically significant secundum atrial septal defect

DETAILED DESCRIPTION:
Prospective, three-stage, single arm, multi-site, clinical investigation evaluating the safety and efficacy of the reSept ASD Occluder in treating clinically significant secundum ASD. Outcomes/endpoints of the clinical investigation will be compared with established performance goals for FDA approved transcatheter secundum ASD occluders.

ELIGIBILITY:
Inclusion Criteria:

All responses must be Yes to be eligible:

1. Age < 85 years.
2. Body weight ≥ 15 kg / 33 lb.
3. Males and Females.
4. Clinically significant, isolated secundum ASD associated with a L-R shunt and signs of RV volume overload that, based upon the expertise of attending physicians requires treatment.
5. ASD of size 5 to 19 mm on screening diagnostic echocardiogram.
6. Isolated secundum ASD of size 8 to 22 mm on stop flow balloon diameter, based upon echocardiographic and fluoroscopic evidence obtained at procedure.
7. Able to take required medications: ASA (Aspirin), low dose (75-100 mg/day), 24 hours prior to and for 6 months following the procedure; Heparin intra-procedurally.
8. Adequate septal rim to support the device. The rim is considered inadequate if it measures less than 5mm in more than two views of a critical structure
9. Adequate defect margin to safely accommodate the selected size implant without interfering with adjacent cardiac structures (e.g., aorta, AV valves, ostia of the pulmonary veins, coronary sinus, or other critical structures), based on the IFU sizing guidance.
10. Capable of giving informed consent, or, for minors, consent of the parent or legal guardian, and willing to comply with the clinical investigation requirements.

Exclusion Criteria:

All responses must be No to be eligible:

1. Pregnancy. Females with child-bearing potential are required to be tested for pregnancy prior to treatment, in accordance with the local institution's policy. For minor females, a pregnancy test will be done in accordance with the local institution's policy.
2. Any significant valve dysfunction that contraindicates ASD closure, or increased pulmonary vascular resistance/severe pulmonary hypertension.
3. Acquired pathological or congenital abnormalities of the cardiovascular system (other than isolated secundum ASD; e.g. congenital malformations, calcification, myocardial infarction, intracardiac thrombi, dilated cardiomyopathy, untreated coronary disease or CAD treated with a stent in the prior 12 months) being clinically significant, that would interfere with the conduct of the clinical investigation.
4. Subjects having undergone left sided structural heart interventions performed via transseptal access (e.g. Mitraclip, LAAO, percutaneous mitral valve replacement).
5. Evidence of thrombus in the left atrium, left atrial appendage, other cardiac chamber, or the inferior vena cava.
6. Sepsis or any other infection that was not successfully treated at least 30 days prior to device placement.
7. Active endocarditis or other infection(s) producing bacteremia.
8. History of atrial tachycardia, atrial fibrillation or flutter, AV block, or ventricular arrhythmia requiring antiarrhythmic medication, pacemaker or AICD.
9. Vasculature is of inadequate size to accommodate all procedural instrumentation.
10. Known allergy to investigational device components or medications, or other contraindication to clinical investigation medications (acetylsalicylic acid, heparin), including a documented history of bleeding, clotting or coagulation disorders, untreated ulcer or any other contraindications to acetylsalicylic acid or antiplatelet therapy.
11. Known hypercoagulable state.
12. Any disorder in the investigator's opinion that could interfere with compliance of safety evaluation as well as any severe concurrent illness that would limit life expectancy (e.g. malignancies).
13. Currently an active subject in an investigational drug or device study that could confound the results of this study.
14. Patients who, in the opinion of the investigator, are inappropriate for inclusion into this clinical investigation or will not comply with requirements of the clinical investigation.
15. Are known to abuse drugs or alcohol.
16. Patients with the diagnosis of Patent Foramen Ovale (PFO).

Max Age: 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with 12-Month Composite Clinical Success | 12 months
  1. Clinically effective ASD closure, defined as no residual ASD or clinically insignificant residual ASD as determined by core laboratory review; and
  2. No re-intervention to treat the defect; and
  3. No device or procedure related serious adverse event.
Number of Subjects with CEC adjudicated Device- or Procedure-related SAEs | 12 months
  Incidence of subjects experiencing one or more serious device- or procedure related adverse events through the 12 month follow up visit, as adjudicated by the Clinical Events Committee (CEC)

SECONDARY OUTCOMES:
ASD Closure Success among Technical Success Subjects | 1 month, 6 months and 12 months
  Assessment of device performance will include closure success, among subjects that were technical successes (i.e. successful placement and release of the reSept ASD Occluder at the ASD), defined as no residual ASD or clinically insignificant residual ASD determined by echocardiography. Assessment of closure success at each follow up through the 12-month follow up will be assessed by TTE.
Number of Subjects with Device- or Procedure-related AEs | 12 months
  Incidence of subjects experiencing one or more non serious device- or procedure-related adverse events through the 12-month follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forbes, MD, Principal Investigator — Joe DiMaggio Children's Hospital/Memorial Healthcare; Saibal Kar, MD, Principal Investigator — Los Robles Regional Medical Center
Locations (32):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Joe DiMaggio Children's Hospital/Memorial Healthcare System, Hollywood, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Toronto General Hospital, Toronto, Canada
- France (5):
  - Hôpital cardiologique Haut-Leveque (CHU Bordeaux), Bordeaux
  - Service de Cardiologie Pédiatrique et Congénitale, Lille
  - Hôpital Mere Enfants (CHU Nantes), Nantes
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital des Enfants (CHU Toulouse), Toulouse
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No